CLINICAL TRIAL: NCT01440790
Title: The Effect of Continuous Sipping of a Glucose Solution on Markers of Oxidation in Men and Women
Acronym: AOGI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Thomas Wolever, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 25401TW
Record Dates: First submitted 2011-08-03; First posted 2011-09-27 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Cardiovascular Disease; Diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Glucose bolus alone (Placebo Comparator): 50g glucose dissolved in water and consumed within 5 minutes.
  Interventions: Dietary Supplement: glucose bolus
- Glucose sipping alone (Experimental): 50g glucose dissolved in water and consumed gradually over 3 hours.
  Interventions: Dietary Supplement: Glucose sipping
- Glucose bolus plus 1g vitamin C (Active Comparator): 50g glucose dissolved in water and consumed in 5 minutes with 1g vitamin C
  Interventions: Dietary Supplement: Glucose bolus plus 1g vitamin C
- Glucose sipping plus 1g vitamin C (Experimental): 50g glucose dissolved in water and consumed gradually of 3 hours. In addition 1g vitamin C will be taken with the first mouthful of glucose solution.
  Interventions: Dietary Supplement: Glucose sipping plus 1g vitamin C

INTERVENTIONS:
Dietary Supplement: glucose bolus — 50g anhydrous glucose dissolved in 300ml water consumed within 10min followed by a lunch (cheese sandwich, fruit and milk) at 4h.
  Arms: Glucose bolus alone
Dietary Supplement: Glucose sipping — 50g anhydrous glucose dissolved in 300ml water consumed at rate of 25ml per 15min followed by a lunch (cheese sandwich, fruit and milk) at 4h.
  Arms: Glucose sipping alone
Dietary Supplement: Glucose bolus plus 1g vitamin C — 50g anhydrous glucose dissolved in 300ml water consumed within 10min with 1g vitamin C followed by a lunch (cheese sandwich, fruit and milk) at 4h.
  Arms: Glucose bolus plus 1g vitamin C
Dietary Supplement: Glucose sipping plus 1g vitamin C — 50g anhydrous glucose dissolved in 300ml water consumed at rate of 25ml per 15min. 1g vitamin C taken with first 25ml. Followed by a lunch (cheese sandwich, fruit and milk) at 4h.
  Arms: Glucose sipping plus 1g vitamin C

SUMMARY:
The objective of this study is to determine the effect of reducing the rate of glucose absorption on oxidative stress after eating and to compare it with the effects of vitamin C. The hypothesis is that reducing the rate of glucose absorption will reduce oxidative stress to a similar extent as 1g vitamin C.

DETAILED DESCRIPTION:
Recently, much attention has been paid to evidence that abnormalities of the postprandial state (hyperglycemia) are important contributing factors to the development of chronic disease. This attention has increased interest in the role low glycemic index (GI) foods could potentially play in preventing postprandial oxidative burst/stress. GI is a means by which to categorize carbohydrate according to their postprandial glycemic response. Low GI foods promote slow intestinal absorption, prolonged and less pronounced postprandial glycemia, may decrease risk of chronic disease, as well as provide metabolic benefit to people living with glucose abnormalities as well as those with normal glucose. Few studies have been conducted looking at the potential relationship between GI and oxidation and are limited by dietary/lifestyle confounders. The proposed study has been developed to eliminate these confounders. Hypotheses (3): 1. Sipping glucose slowly over 3h will result in less oxidative stress than ingesting the same amount of glucose as a bolus over 5min. 2. Sipping glucose will reduce oxidative stress to the same extent as 1g of oral vitamin C. 3. The effect of sipping glucose on oxidative stress will occur sooner than that of vitamin C.

ELIGIBILITY:
Inclusion Criteria:

* healthy males or females
* 18 to 75 years

Exclusion Criteria:

* diabetes
* recent hospitalization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Incremental Area Under the Curve over 4 hours in serum TRAP (total peroxyl radical-trapping potential) | Four (4) hours after starting to eat the test meal.

SECONDARY OUTCOMES:
Change over 6 hours from baseline in Plasma glucose | Baseline and 30, 60, 120, 180, 240, 270, 300 and 360min
Change over 6 hours from baseline in Plasma insulin | Baseline and 30, 60, 120, 180, 240, 270, 300 and 360min
Change over 6 hours from baseline in Plasma free-fatty acids | Baseline and hourly for 6h
Change over 6 hours from baseline in Serum vitamin C | Baseline and 2, 4 and 6h
Change over 6 hours from baseline in C-reactive protein | Baseline and 2, 4 and 6h
Change over 6 hours from baseline in Blood pressure | Baseline and 1, 2, 4, 5 and 6h
Change over 6 hours from baseline in Pulse | Baseline and 1, 2, 4, 5 and 6h
Change over 6 hours from baseline in Pulse pressure | Baseline and 1, 2, 4, 5 and 6h
Change over 6 hours from baseline in Augmentation index | Baseline and 1, 2, 4, 5 and 6h
Change over 6 hours from baseline in Oxidized LDL | Baseline and hourly for 6hr
Change from baseline in serum TRAP over 6 hours | Baseline and 30, 60, 120, 180, 240, 270, 300 and 360min

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, BMBCh PhD DM, Principal Investigator — University of Toronto; Shannan Grant, MSc, RD, Study Director — University of Toronto